CLINICAL TRIAL: NCT06687018
Title: Comparative Effects of Kaltenborn Versus Mulligan Mobilisation on Pain, Disability and Hand Function in Patients With Carpal Tunnel Syndrome
Brief Title: Effects of Kaltenborn and Mulligan Mobilisation in Patients With Carpal Tunnel Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0129
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Kaltenborn, Mulligan, Pain, Disability, Hand Function, CTS
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaltenborn mobilisation (Experimental): Kaltenborn mobilisation along with conventional treatment.
  Interventions: Other: Kaltenborn mobilisation
- Mulligan mobilisation (Active Comparator): Mulligan mobilisation along with conventional treatment.
  Interventions: Other: Mulligan mobilisation

INTERVENTIONS:
Other: Kaltenborn mobilisation — Kaltenborn mobilisation Grade 3 along with common treatment for 3 minutes, repeated 3 sets with rest of 1 minutes, three sessions per week for four weeks. Conventional treatment comprises a hot pack for 10 minutes, SWD for 5 minutes, and nerve and tendon gliding exercises.
  Arms: Kaltenborn mobilisation
Other: Mulligan mobilisation — Mulligan mobilisation with 10 repetitions with 3 sets and three sessions per week for four weeks. Conventional treatment comprises a hot pack for 10 minutes, SWD for 5 minutes, and nerve and tendon gliding exercises
  Arms: Mulligan mobilisation

SUMMARY:
Carpal Tunnel Syndrome is the most common mononeuropathy that results from the compression of median nerve in carpal tunnel, leading to entrapment neuropathy. The symptoms become aggravated during drawing, typing or playing video games. The aim of study will be to compare the effects of Kaltenborn and Mulligan mobilisation on pain, disability and hand function in patients with carpal tunnel syndrome.

DETAILED DESCRIPTION:
This research will adopt a Randomized Clinical Trial design. Upon approval of the synopsis, ethical clearance would be taken and necessary permissions from Ejaz Hospital Lahore. Through convenience sampling technique, 48 patients will be included which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Mobilisation technique includes moving the proximal row of carpal bones either dorsally to promote wrist extension or to the palmar side to promote wrist flexion. Group A will be treated with Grade 3 Kaltenborn mobilisation. Grade 3 distraction was chosen to avoid contact between the articular surfaces and to stimulate hypoalgesic factors and Group B will be treated with Mulligan mobilisation. Outcome measures will be conducted through pain, disability and hand function questionnaire after 6 weeks. Data will be analyzed during SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Both genders between 20 and 45 years of age
* Individuals having localized pain, tingling and numbness in the median nerve distribution
* Positive Tinel sign and positive Phalen's test

Exclusion Criteria:

* Any sensory and/or motor deficit in either the ulnar or radial nerve traumatic neck injury
* Previous hand surgery or trauma or cervical radiculopathy
* Systemic disease e.g. diabetes mellitus or thyroid disease or rheumatoid arthritis

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  Changes from baseline, Numeric Rating Scale (NRS) is the most commonly used scale in which the pain rate ranges from 0 (no pain) to 10 (worst pain). The NPRS has validity of 0.86 to 0.95 and reliability of 0.96.
Boston Carpal Tunnel Questionnaire | 4 weeks
  Questionnaire used to assess functional status and symptom severity. There are two subscales in BCTQ. The Functional Status Scale evaluates hand function, whereas the Symptom Severity Scale (SSS) provides PRO data on the degree of symptoms. Eleven items make up the Symptom Severity scale, which rates symptoms related to pain, paresthesia, numbness, weakness, and grasping trouble. Eight items make up the Functional Status Scale (FSS), which evaluates functional deficiencies. Form 1 (no symptoms/difficulties) to 5 (worst symptoms/cannot do the task at all) each item is graded.(20). In BCQT, SSS has reliability 0.89 and FSS has 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Ejaz Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bougea A, Zambelis T, Voskou P, Katsika PZ, Tzavara C, Kokotis P, Karandreas N. Reliability and Validation of the Greek Version of the Boston Carpal Tunnel Questionnaire. Hand (N Y). 2018 Sep;13(5):593-599. doi: 10.1177/1558944717725379. Epub 2017 Aug 20. PMID 28825339
- [Background] Abdolrazaghi HA, Khansari M, Mirshahi M, Ahmadi Pishkuhi M. Effectiveness of Tendon and Nerve Gliding Exercises in the Treatment of Patients With Mild Idiopathic Carpal Tunnel Syndrome: A Randomized Controlled Trial. Hand (N Y). 2023 Mar;18(2):222-229. doi: 10.1177/15589447211006857. Epub 2021 Apr 15. PMID 33855879
- [Background] Exelby L. Peripheral mobilisations with movement. Man Ther. 1996 Jun;1(3):118-126. doi: 10.1054/math.1996.0259. PMID 11440498
- [Background] Spagnoli AM, Fino P, Fioramonti P, Sanese G, Scuderi N. Bifid median nerve and carpal tunnel syndrome: an uncommon anatomical variation. Ann Ital Chir. 2017;88:95-96. PMID 28447963
- [Background] Li ZM, Jordan DB. Carpal tunnel mechanics and its relevance to carpal tunnel syndrome. Hum Mov Sci. 2023 Feb;87:103044. doi: 10.1016/j.humov.2022.103044. Epub 2022 Nov 25. PMID 36442295
- [Background] Talebi GA, Saadat P, Javadian Y, Taghipour M. Comparison of two manual therapy techniques in patients with carpal tunnel syndrome: A randomized clinical trial. Caspian J Intern Med. 2020;11(2):163-170. doi: 10.22088/cjim.11.2.163. PMID 32509244